CLINICAL TRIAL: NCT02825992
Title: Utilizing Novel Dipole Density Capabilities to Objectively Visualize the Etiology of Rhythms in Atrial Fibrillation (UNCOVER-AF)
Brief Title: Utilizing Novel Dipole Density Capabilities to Objectively Visualize the Etiology of Rhythms in Atrial Fibrillation
Acronym: UNCOVER-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CL-AF-002; CL-AF-001 (Other: Acutus Medical); NCT02462980 (obsolete NCT alias)
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AcQMap System (Other): All patients who underwent catheter ablation using the AcQMap System
  Interventions: Device: AcQMap System

INTERVENTIONS:
Device: AcQMap System — 3D imaging and mapping system for cardiac chambers

SUMMARY:
A prospective, single-arm, multi-center, multi-national, non-randomized, post-market study designed to provide clinical data regarding the use of the AcQMap™ System in the ablation of persistent atrial fibrillation. (CL-AF-002 - EU)

A prospective, single-arm, multi-center, multi-national non-randomized study designed to provide clinical data regarding the use of the AcQMap™ System in the ablation of persistent atrial fibrillation. (CL-AF-001 - Canadian)

DETAILED DESCRIPTION:
A prospective, single-arm, multi-center, multi-national, non-randomized, post-market study designed to provide clinical data regarding the use of the AcQMap™ System in the ablation of persistent atrial fibrillation. (CL-AF-002 - EU)

A prospective, single-arm, multi-center, multi-national non-randomized study designed to provide clinical data regarding the use of the AcQMap™ System in the ablation of persistent atrial fibrillation. (CL-AF-001 - Canadian)

The research study was conducted in the EU and Canada. The protocol and the corresponding NCT number is as follows:

NCT02462980 (Protocol CL-AF-001, Site Ontario, Canada Dr. Verma = PI)

The above record was combined into one as both protocols are essentially identical (one is post market [EU] and the other pre-market [Canada] and one study report will be written that encompasses the data/results for both protocols.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an ablation of persistent atrial fibrillation

Exclusion Criteria:

* Any duration of continuous AF lasting longer than 12 months
* Previous AF ablation
* Significant structural heart disease
* Previous cerebral infarct
* Major bleeding disorders
* Pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Willems, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf (UKE)
Locations (12):
- Southlake Regional Health Center, Newmarket, Ontario, Canada
- Na Homolce Hospital, Prague, Czechia
- Germany (3):
  - Vivantes Klinikum Am Urban, Berlin
  - Herzzentrum der Universität zu Köln, Cologne
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Centro Cardiologico Monzino, Milan, Italy
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - St. Antonius Hospital, Nieuwegein
- United Kingdom (4):
  - Freeman Hospital, Newcastle, Newcastle Upon Tyne
  - Papworth Hospital, Cambridge
  - Royal Brompton Hospital, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Willems S, Verma A, Betts TR, Murray S, Neuzil P, Ince H, Steven D, Sultan A, Heck PM, Hall MC, Tondo C, Pison L, Wong T, Boersma LV, Meyer C, Grace A. Targeting Nonpulmonary Vein Sources in Persistent Atrial Fibrillation Identified by Noncontact Charge Density Mapping: UNCOVER AF Trial. Circ Arrhythm Electrophysiol. 2019 Jul;12(7):e007233. doi: 10.1161/CIRCEP.119.007233. Epub 2019 Jun 27. PMID 31242746

RESULTS

PARTICIPANT FLOW:
Groups:
- AcQMap System: Use of the AcQMap System for imaging and mapping of atrial chambers during AF ablation
  AcQMap System: 3D imaging and mapping system for cardiac chambers
Period: Overall Study
Arm/Group | AcQMap System
Started | 129 (The procedure was terminated for clinical reasons in 2 patients, therefore only 127 were treated.)
Completed | 121
Not Completed | 8
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 2
Not completed — Procedure terminated | 2

BASELINE CHARACTERISTICS:
Arm/Group | AcQMap System
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 128
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 129
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4
  Netherlands | 8
  Czechia | 11
  United Kingdom | 54
  Italy | 6
  Germany | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From Device/Procedure Related Major Adverse Events (MAEs)
Description: MAEs include: Death, cardiac perforation, cerebral infarct, systemic embolism, major bleeding, cardiac valve damage.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | AcQMap System
Number analyzed (Participants) | 129
Participants
  Number of subjects with MAEs | 3
  Number of subjects with no MAEs | 126

2. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Events.
Description: Recording of all adverse events through 12 month follow-up
Time Frame: 12 Months
Population: The safety population included all enrolled subjects who had the venous access portion of the ablation procedure initiated.
Measure: Number; unit: participants
Arm/Group | AcQMap System
Number analyzed (Participants) | 129
participants
  ERYTHEMA OF EXTREMITIES | 1
  BLOOD AND LYMPHATIC SYSTEM DISORDERS | 1
  CARDIAC DISORDERS | 21
  CONGENITAL, FAMILIAL AND GENETIC DISORDERS | 1
  ENDOCRINE DISORDERS | 3
  EYE DISORDERS | 1
  GASTROINTESTINAL DISORDERS | 8
  GENERAL DISORDERS AND ADMIN SITE CONDITIONS | 17
  HEPATOBILIARY DISORDERS | 2
  INFECTIONS AND INFESTATIONS | 11
  INJURY, POISONING AND PROCEDURAL COMPLICATIONS | 6
  INVESTIGATIONS | 6
  METABOLISM AND NUTRITION DISORDERS | 2
  MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS | 2
  NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED | 4
  NERVOUS SYSTEM DISORDERS | 7
  PSYCHIATRIC DISORDERS | 1
  RENAL AND URINARY DISORDERS | 5
  RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS | 10
  SKIN AND SUBCUTANEOUS TISSUE DISORDERS | 1
  SURGICAL AND MEDICAL PROCEDURES | 3
  VASCULAR DISORDERS | 16

3. Secondary Outcome: Number of Participants Who Were in Sinus Rhythm Following the Ablation Procedure.
Description: Conversion to sinus rhythm post ablation
Time Frame: 24 hours
Population: Number of subjects who had an ablation procedure completed
Measure: Count of Participants; unit: Participants
Arm/Group | AcQMap System
Number analyzed (Participants) | 127
Participants | 125

4. Secondary Outcome: Number of Participants Who Were AF Free at, 6, 9, and 12 Months Post Ablation.
Description: Freedom from AF
Time Frame: 6, 9, and 12 Months
Measure: Count of Participants; unit: Participants
Groups:
- 6 Month Off AADs: Freedom from AF at 6 Months post ablation off Anti-Arrhythmic Drug (AADs)
- 6 Month on AADs: Freedom from AF at 6 Months post ablation on Anti-Arrhythmic Drug (AADs)
- 9 Months Off AADs: Freedom from AF at 9 Months post ablation off Anti-Arrhythmic Drug (AADs)
- 9 Months on AADs: Freedom from AF at 9 Months post ablation on Anti-Arrhythmic Drug (AADs)
- 12 Months Off AADs: Freedom from AF at 12 Months post ablation off Anti-Arrhythmic Drug (AADs)
- 12 Months on AADs: Freedom from AF at 12 Months post ablation on Anti-Arrhythmic Drug (AADs)
Arm/Group | 6 Month Off AADs | 6 Month on AADs | 9 Months Off AADs | 9 Months on AADs | 12 Months Off AADs | 12 Months on AADs
Number analyzed (Participants) | 112 | 112 | 88 | 88 | 118 | 118
Participants | 79 | 49 | 65 | 36 | 84 | 52

ADVERSE EVENTS:
Time Frame: Adverse Events were collected through 12 months post-procedure.
Arm/Group | AcQMap System
All-Cause Mortality (participants affected / at risk) | 0/129
Serious Adverse Events (participants affected / at risk) | 33/129
Other Adverse Events (participants affected / at risk) | 58/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AcQMap System (N=129)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 2 (2)
ATRIAL TACHYCARDIA (Cardiac disorders) | 2 (2)
BRADYCARDIA (Cardiac disorders) | 2 (2)
CARDIAC FAILURE (Cardiac disorders) | 2 (2)
PNEUMONIA (Infections and infestations) | 3 (3)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 2 (3)
ARTERIOVENOUS FISTULA (Vascular disorders) | 3 (3)
HYPOTENSION (Vascular disorders) | 2 (2)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
CARDIAC TAMPONADE (Cardiac disorders) | 1 (1)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 (1)
SINUS ARREST (Cardiac disorders) | 1 (1)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
CHEST DISCOMFORT (General disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
INFLAMMATION (General disorders) | 1 (1)
JAUNDICE (Hepatobiliary disorders) | 1 (1)
ARTERIOGRAM CORONARY (Investigations) | 1 (1)
CATHETERISATION CARDIAC (Investigations) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 1 (1)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NEOPLASM RECURRENCE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (3)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY MASS (Reproductive system and breast disorders) | 1 (1)
ABDOMINAL HERNIA REPAIR (Surgical and medical procedures) | 1 (1)
LYMPHOCELE (Vascular disorders) | 1 (1)
PERICARDIAL EFFUSION (Congenital, familial and genetic disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AcQMap System (N=129)
ANGINA PECTORIS (Cardiac disorders) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 2 (2)
HYPERTHYROIDISM (Endocrine disorders) | 3 (3)
CHEST PAIN (General disorders) | 3 (3)
FATIGUE (General disorders) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 6 (6)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2)
PNEUMONIA (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 (5)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ARTERIOVENOUS FISTULA (Vascular disorders) | 2 (2)
HAEMATOMA (Vascular disorders) | 6 (6)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 (1)
INTRACARDIAC THROMBUS (Cardiac disorders) | 1 (1)
PERICARDITIS (Cardiac disorders) | 1 (1)
BLINDNESS TRANSIENT (Eye disorders) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 (1)
TOOTH SOCKET HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
ADMINISTRATION SITE ERYTHEMA (General disorders) | 2 (2)
CHILLS (General disorders) | 1 (1)
OEDEMA (General disorders) | 1 (1)
PUNCTURE SITE HAEMORRHAGE (General disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
VASCULAR ACCESS SITE RUPTURE (Injury, poisoning and procedural complications) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1)
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 1 (1)
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
GOUT (Metabolism and nutrition disorders) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ATYPICAL FIBROXANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 (1)
CARDIAC ABLATION (Surgical and medical procedures) | 1 (1)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 1 (1)
AIR EMBOLISM (Vascular disorders) | 1 (1)
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
PHLEBITIS (Vascular disorders) | 1 (1)
ERYTHEMA OF EXTREMITIES (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Identified limitations

* Not an RCT limiting the comparability of the results to current SOC
* A first-generation device study with limited experienced users. Outcome measures may not be reflective of current clinical results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
None of the results, in whole or part, of the study carried out under the study protocol, nor any of the information provided by the sponsor for the purposes of performing the study, were allowed to be published or passed on to any third party without the consent of the sponsor. Any Investigator involved with this study was obligated to provide the sponsor with complete test results and all data derived from the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT02825992/Prot_SAP_000.pdf